CLINICAL TRIAL: NCT00089778
Title: Immunization of Patients With Renal Cancer Using HLA-A2 and HLA-A3-Binding Peptides From Fibroblast Growth Factors 5 (FGF-5)
Brief Title: Vaccine Treatment of Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: fewer tumors than expected expressed FGF-5, led to end of accrual to cohorts A&B
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Yang, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 040259; 04-C-0259; NCT00091403 (obsolete NCT alias)
Record Dates: First submitted 2004-08-12; First posted 2004-08-13 (Estimated); Results first posted 2012-10-11 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Kidney Cancer
Keywords: Clinical Response; Toxicity; Immunologic Response; Adjuvant; IL-2; Renal Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Fibroblast Growth Factor 5; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Grp A-Measurable metastatic disease (no immediate aldesleukin) (Experimental): Patients who do not need or are ineligible for treatment with interleukin-2 (IL-2) and patients who have previously had IL-2 therapy.
  A3 FGF-5 (Fibroblast growth factor 5): 172-176/217-220 peptide - two 1 ml injections in the anterior thigh deep subcutaneous tissue within 2c of each other.
  Interventions: Drug: Fibroblast growth factor 5 (FGF-5):172-176/217-220
- Grp B - Measurable metastatic disease that require aldesleukin (Experimental): Patients who require immediate treatment with IL-2. A2 FGF-5: 117-126 peptide + HD (high dose) IL-2 (prior cycle 1)- two 1 ml injection in the anterior thigh deep subcutaneous tissue within 2c of each other.
  720,000 IU/kg as an intravenous bolus over a 15 minute period every 8 hours beginning on the day after immunization and continuing for up to 4 days (a maximum of 12 doses).
  Interventions: Drug: 117-126:Fibroblast growth factor 5 (FGF-5); Other: IL-2
- Grp C - High-risk loco-regional disease (Experimental): Patients whose cancer has been surgically removed but who are at risk for recurrence and local disease and who are seeking experimental adjuvant therapy.
  A2 FGF-5: 117-126 peptide (adjuvant); A3 FGF-5: 172-176/217-220 peptide (adjuvant)
  Interventions: Drug: 117-126:Fibroblast growth factor 5 (FGF-5)

INTERVENTIONS:
Drug: 117-126:Fibroblast growth factor 5 (FGF-5) — Two 1 ml injection in the anterior thigh deep subcutaneous tissue within 2c of each other.
  Other Names: MLSVLEIFAV
  Arms: Grp B - Measurable metastatic disease that require aldesleukin; Grp C - High-risk loco-regional disease
Drug: Fibroblast growth factor 5 (FGF-5):172-176/217-220 — Two 1 ml injection in the anterior thigh deep subcutaneous tissue within 2c of each other.
  Other Names: NTYASPRFK
  Arms: Grp A-Measurable metastatic disease (no immediate aldesleukin)
Other: IL-2 — 720,000 IU/kg as an intravenous bolus over a 15 minute period every 8 hours beginning on the day after immunization and continuing for up to 4 days (a maximum of 12 doses).
  Other Names: Interleukin-2; Aldesleukin
  Arms: Grp B - Measurable metastatic disease that require aldesleukin

SUMMARY:
This study will evaluate the safety and side effects of two experimental vaccines in patients with kidney cancer and determine whether the vaccines "turn on" an immune response to the cancer. Each vaccine contains one of two peptides (pieces of proteins) from the fibroblast growth factor 5 (FGF-5) antigen, a protein produced by some cancer cells, and an oil-based liquid called Incomplete Freud's Adjuvant (Montanide ISA-51) that enhances the immune response to the vaccine.

Patients 16 years of age and older who have kidney cancer that has spread beyond the kidney or whose primary kidney tumor has been removed within 6 months before entering the study and are at high risk for disease recurrence may be eligible for this study. Patients must have tissue type human leukocyte antigen serotype within HLA-A A serotype group (HLA-A2) or human leukocyte antigen serotype within HLA-A A serotype group (HLA-A3) (determined by a blood test for human leukocyte antigen (HLA) typing) and their tumors must produce the FGF-5 peptide. Candidates are screened with a physical examination, blood and urine tests, electrocardiogram (EKG), tumor biopsy (removal of a small sample of tumor for examination) in patients whose tumor is easily accessible, and scans (computed tomography (CT), bone scans) and x-rays if current scans are not available.

Participants are divided into two groups according to their HLA type (HLA-A2 or HLA-A3) to receive the vaccine appropriate for their HLA type. They are then further divided into three groups: 1) Group 1 includes patients who do not need or are ineligible for treatment with interleukin-2 (IL-2), a protein made by certain infection-fighting white cells that helps fight tumors) and patients who have previously had IL-2 therapy; 2) Group 2 includes patients who require immediate treatment with IL-2; and 3) Group 3 includes patients whose cancer has been surgically removed but who are at risk for recurrence.

Patients in Groups 1 and 3 receive two peptide injections four times a week every 3 weeks for up to a year, or until their tumor grows (or returns in patients in Group 3) or the side effects are too severe to continue. Tumors are evaluated with a physical examination and scans or x-rays every 12 weeks and blood tests are done every 3 weeks. Patients in Group 2 receive two peptide injections every day for 4 days, along with doses of IL-2 starting the day after the first peptide injection. The vaccines are given as injections under the skin of the thigh. IL-2 is infused through a vein over 15 minutes every 8 hours for up to 12 doses, depending on tolerance. The vaccine and IL-2 are repeated every 10 to 14 days, with tumor evaluations every 2 months. Patients stay in the hospital about 1 week during each treatment cycle to receive the IL-2.

All patients undergo leukapheresis, a procedure for collecting large numbers of white blood cells. Blood is collected through a needle in an arm vein and flows through a cell separator machine, where the white cells are extracted. The rest of the blood is returned to the patient through the same needle or a needle in the other arm. The white cells are examined to evaluate how the vaccines change the action of immune cells. Some patients may undergo an additional biopsy of normal skin and tumor or lymph node to look at the effects of the vaccine on the immune cells in the tumor.

Patients in Group 1 whose cancer grows and patients in Group C whose cancer returns may be offered IL-2 treatments as given to Group 2 patients, along with the peptide vaccine. If the disease responds to IL-2, the treatment may be repeated after 2 months.

DETAILED DESCRIPTION:
Background:

Several preliminary clinical results in the treatment of cancer lend credence to the hypothesis that augmented T-cell responses will improve IL-2 therapy. A peptide vaccine derived from the melanoma/melanosomal antigen, GP100, when given with high-dose IL-2 resulted in a response rate over 30% in a small Phase II study. These results have led to efforts to identify similar T-cells and tumor-associated antigens for IL-2 responsive tumors such as renal cell cancer. Work in our laboratory generated a renal cancer-reactive T-cell clone, raised from tumor-infiltrating lymphocytes (TIL) within a renal cell cancer (RCC) metastasis undergoing spontaneous regression. This clone was HLA-A3 restricted and recognized autologous tumor as well as a number of allogeneic RCC lines also expressing HLA-A3. Expression cloning of the antigen recognized by this clone demonstrated that the RCC-associated antigen being recognized was unmutated fibroblast growth factor 5 (FGF-5). We concluded from numerous studies that FGF-5 was a tumor associated antigen over-expressed by a majority of RCC and that it had several favorable characteristics as a target for immunotherapy. At this point, having demonstrated in the laboratory that tumor-reactive T-cells generated from patients with renal cancer can recognize naturally presented FGF-5 in either the context of HLA-A2 or HLA-A3 via the minimal determinants 117-126:FGF-5 (MLSVLEIFAV) or FGF-5:172-176/217-220 (NTYASPRFK), respectively. With this study we plan to determine if vaccination with these peptides can enhance the number of FGF-5-reactive cytotoxic T lymphocytes (CTL) precursors in patients with renal cancer or affect the anticipated response rate from high-dose IL-2.

Objectives:

The primary objective for patients with renal cell carcinoma will be to determine overall response rates and toxicity of peptide vaccination with HLA-A2 and HLA-A3- binding peptides from FGF-5 in HLA-appropriate patients, and to explore the effect of such vaccination on the response rate to high-dose IL-2. The primary objective for patients who are receiving vaccination in the adjuvant setting will be to evaluate the immunologic responses and toxicity of FGF-5 peptide vaccination who are likely to receive repeat vaccination prior to requiring IL-2. The secondary objective is to evaluate the immunologic responses to FGF-5 peptide vaccination.

Eligibility:

Patients who are HLA-A2+ or HLA-A3+, must be age greater than or equal to 16, and have an expected survival greater than three months. For cohort A and B, patients must have measurable metastatic renal cancer and FGF-5 tumor expression. For cohort C, patients are required to have had a Stage III primary tumor (i.e. T3/T4 or N1/N2) excised within the last 6 months.) Patients in cohorts A and B must have tumor sites safely accessible for biopsy or indications for resection of a site of tumor (e.g. an indicated nephrectomy or symptomatic metastasis) and be willing to undergo biopsy, and have FGF-5 expression determined by reverse transcription polymerase chain reaction (RT-PCR) and will only be eligible if it is detectable. Patients must meet specific safety laboratory criteria. May not have undergone other systemic therapies for their cancer in the past 3 weeks (6 weeks for nitrosureas), not have any major medical illnesses, or require systemic steroid therapy.

Design:

Patients will first be divided into cohorts with measurable metastatic disease (Cohorts A and B) or high-risk loco-regional disease (Cohort C). Patients with measurable metastatic disease will then be separated into those who require immediate IL-2 therapy (Cohort B) or those who do not (cohort A).

Cohort A will begin receiving vaccination with HLA-appropriate peptide emulsified in Montanide ISA-51 or Montanide® (Registered Trademark) ISA 51 VG daily for four days every 3 weeks and will continue this for up to a year, or until tumor progression is documented. At that point, those ineligible for high-dose IL-2 or who have had previous IL-2 as an inpatient (considered high dose at doses greater than or equal to 600,000 IU/kg) will be taken off of study, and those still eligible for IL-2 who have not yet received it, will have high-dose intravenous bolus IL-2 (720,000 IU/kg/dose every 8 hours up to 12 doses) added to their peptide vaccination regimen. Two cycles, separated by 10-14 days, will be given during every two-month period (constitutes a course.). Patients in Cohort A crossing over to vaccination plus IL-2 therapy, will receive peptide in MONTANIDE ISA-51 or Montanide® (Registered Trademark) ISA 51 VG vaccination the day prior to starting an IL-2 cycle (instead of every 3 weeks, to accommodate the IL-2 regimen) and repeated daily for three additional days (for a total of four days) during IL-2 administration.

Patients in Cohort B will begin with high-dose bolus IL-2 therapy in two cycles within every two month period, with each cycle preceded by a peptide in MONTANIDE ISA-51 or Montanide® (Registered Trademark) ISA 51 VG vaccine the day prior to starting each IL-2 cycle with peptide in MONTANIDE ISA-51 or Montanide® (Registered Trademark) ISA 51 VG repeated daily for three additional days (for a total of four days) during IL-2 administration.

Patients in Cohort C will undergo the same HLA-appropriate vaccination with peptide and MONTANIDE ISA-51 or Montanide® (Registered Trademark) ISA 51 VG daily for four days every 3 weeks and continue for up to 6 months or until disease relapse is documented. At the time of relapse, eligible patients in Cohort C will receive treatment with high-dose bolus IL-2 and continuing peptide vaccination using the same schedule as specified for the Cohort A crossover arm above.

For patients in cohort A on peptide vaccine alone, evaluation will be performed every 3 months during the first 6 months of therapy and if stable, every 3-6 months thereafter. For cohorts A and B during peptide vaccine plus high-dose IL-2 therapy, evaluation will be performed every 2 months while on IL-2, and every 3-6 months for stable patients off therapy. For cohort C, evaluations will be performed every 3 months for the first year and every 6-12 months thereafter.

The maximal accrual possible would be 210 patients (Cohort A with 80 patients, Cohort B with 66 patients and Cohort C with 64 patients), and maximal enrollment could take up to 5 years.

ELIGIBILITY:
* INCLUSION CRITERIA

Patients will be screened for inclusion on this study while participating in the Surgery Branch protocol 99-C-0128: Evaluation for the National Cancer Institute (NCI) Surgery Branch Clinical Research Protocols

Patients with clear cell renal carcinoma must fall into one of the two following groups:

For cohort A and B, patients must have measurable metastatic renal cancer and fibroblast growth factor 5 (FGF-5) tumor expression. For cohort C, patients are required to have had a Stage III primary tumor (i.e. T3/T4 or N1/N2) excised within the last 6 months.

Patients must be greater than or equal to 16.

Expected survival must be greater than three months

Patients in cohorts A and B must have tumor sites safely accessible for biopsy or indications for resection of a site of tumor (e.g. an indicated nephrectomy or symptomatic metastasis) and have FGF-5 expression determined by RT-PCR (reverse transcription polymerase chain reaction) and will only be eligible if it is detectable.

Must be human leukocyte antigen serotype within HLA-A A serotype group (HLA-A2+) or HLA-A3+.

Serum creatinine of 2.0 mg/dl or less.

Bilirubin 1.6 mg/dl or less, except in patients with Gilbert's syndrome who must have a total bilirubin less than 3.0 mg/dl.

White blood cell (WBC) 3000/mm or greater.

Platelet count 90,000mm^3 or greater.

Serum aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less then three times normal.

Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Patients of both genders must be willing to practice effective birth control during this trial and for three months after active treatment on this trial.

Patients who have received previous low dose interleukin-2 (IL-2) (less than 600,000 IU/kg Food and Drug Administration (FDA) approved dosing regimen) will be eligible.

For cohort A for each human leukocyte antigen (HLA) type, if there are no clinical responses to vaccine alone in the first 12 patients enrolled, subsequent patients must be eligible to receive high-dose IL-2.

Patients must be able to understand and sign the informed consent document.

Eligibility for administration of IL-2.

Patients must meet the following criteria to be eligible to receive IL-2:

Patients may not have active major medical illnesses such as cardiac ischemia, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.

Patients with recent prolonged history of cigarette smoking or symptoms of respiratory dysfunction must have a normal pulmonary function test as evidenced by a forced expiratory volume in 1 second (FEV1) greater than 60% predicted.

Patients with electrocardiogram (EKG) abnormalities, symptoms of cardiac ischemia or arrhythmias or age greater than 50 years will have a normal stress cardiac test (stress thallium, stress multi-gated acquisition scan (MUGA), dobutamine echocardiogram or other stress test).

Patients must be willing to sign a durable power of attorney (DPA).

Serum creatinine of 2.0 mg/dl or less.

Total bilirubin 2.0 mg/dl or less, except in patients with Gilbert's syndrome who must have a total bilirubin less than 3.0 mg/dl.

White blood cell (WBC) 3000/mm^3 or greater.

Platelet count 90,000 mm^3 or greater.

EXCLUSION CRITERIA:

Patients will be excluded:

Who are not willing or able to be biopsied.

Who are undergoing or have undergone in the past 3 weeks any other form of therapy for their cancer, or have undergone nitrosurea therapy within the past 6 weeks. All patients toxicities must have recovered to a grade 1 or less. Patients may have undergone minor surgical procedures or local radiotherapy within the past 3 weeks as long as all toxicities have recovered to a grade 1 or less.

Have active systemic infections, coagulation disorder, or other major medical illnesses of the cardiovascular or respiratory symptoms or any known immunodeficiency disease (Immune competence will be defined as lymphocyte count greater than 500 (grade 3 toxicity in Common Toxicity Criteria (CTC) 3); white blood cell (WBC) 1000; and absence of opportunistic infections).

Who require systemic steroid therapy.

Who are pregnant (because of possible side effects on the fetus) or who are breastfeeding, or who are unwilling/unable to practice effective birth control.

Who are known to be positive for hepatitis BsAG, or human immunodeficiency virus (HIV) antibody, or hepatitis C antibody (unless antigen negative), (because of possible immune effects of these conditions).

Who have had a known allergic reaction to Incomplete Freund's Adjuvant (MONTANIDE ISA-51) or hypersensitivity to any agent used on this protocol.

Who have a fresh tumor specimen with no evidence of FGF-5 expression on a technically adequate RT-PCR assessment.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2004-09-10 (Actual); Primary Completion 2008-08-05 (Actual); Study Completion 2008-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Yang, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Bruggen P, Traversari C, Chomez P, Lurquin C, De Plaen E, Van den Eynde B, Knuth A, Boon T. A gene encoding an antigen recognized by cytolytic T lymphocytes on a human melanoma. Science. 1991 Dec 13;254(5038):1643-7. doi: 10.1126/science.1840703.
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/A_2004-C-0259.html
- See also: Common Toxicity Criteria version 3.0 (CTCv3) — http://ctep.cancer.gov

RESULTS

PARTICIPANT FLOW:
Groups:
- Grp A-measurable Metastatic Disease (no Immediate Aldesleukin): Patients who do not need or are ineligible for treatment with interleukin-2 (IL-2) and patients who have previously had IL-2 therapy.
  A3 FGF-5 (Fibroblast growth factor 5): 172-176/217-220 peptide - two 1 ml injections in the anterior thigh deep subcutaneous tissue within 2c of each other.
  This is not a conventional crossover-If a patient in Group C has a recurrence after vaccination or cancer progresses in Group A, then we wanted to administer an approved, conventional therapy for recurrent disease (IL-2) which could have had synergy with the prior experimental vaccination. This was only exploratory and there was no specific endpoint targeted in patient's crossing over and there was no impact on study size (too involved for the scope of this study).
- Grp B - Measurable Metastatic Disease That Require Aldesleukin: Patients who require immediate treatment with IL-2. A2 FGF-5: 117-126 peptide + HD (high dose) IL-2 (prior cycle 1) Two 1 ml injection in the anterior thigh deep subcutaneous tissue within 2c of each other.
  720,000 IU/kg as an intravenous bolus over a 15 minute period every 8 hours beginning on the day after immunization and continuing for up to 4 days (a maximum of 12 doses).
  This is not a conventional crossover-If a patient in Group C has a recurrence after vaccination or cancer progresses in Group A, then we wanted to administer an approved, conventional therapy for recurrent disease (IL-2) which could have had synergy with the prior experimental vaccination. This was only exploratory and there was no specific endpoint targeted in patient's crossing over and there was no impact on study size (too involved for the scope of this study).
- Grp C - High-risk Loco-regional Disease: Patients whose cancer has been surgically removed but who are at risk for recurrence and local disease and who are seeking experimental adjuvant therapy.
  A2 FGF-5: 117-126 peptide (adjuvant); A3 FGF-5: 172-176/217-220 peptide (adjuvant).
  This is not a conventional crossover-If a patient in Group C has a recurrence after vaccination or cancer progresses in Group A, then we wanted to administer an approved, conventional therapy for recurrent disease (IL-2) which could have had synergy with the prior experimental vaccination. This was only exploratory and there was no specific endpoint targeted in patient's crossing over and there was no impact on study size (too involved for the scope of this study).
Period: Overall Study
Arm/Group | Grp A-measurable Metastatic Disease (no Immediate Aldesleukin) | Grp B - Measurable Metastatic Disease That Require Aldesleukin | Grp C - High-risk Loco-regional Disease
Started | 2 | 1 | 8
Completed | 2 | 1 | 7
Not Completed | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Grp B - Measurable Metastatic Disease That Require Aldesleukin: Patients who require immediate treatment with IL-2. A2 FGF-5: 117-126 peptide + HD (high dose) IL-2 (prior cycle 1) Two 1 ml injection in the anterior thigh deep subcutaneous tissue within 2c of each other.
  720,000 IU/kg as an intravenous bolus over a 15 minute period every 8 hours beginning on the day after immunization and continuing for up to 4 days (a maximum of 12 doses).
- Total: Total of all reporting groups
Arm/Group | Grp A-measurable Metastatic Disease (no Immediate Aldesleukin) | Grp B - Measurable Metastatic Disease That Require Aldesleukin | Grp C - High-risk Loco-regional Disease | Total
Number analyzed (Participants) | 2 | 1 | 8 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 7 | 10
  >=65 years | 0 | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (2.8) | 54.0 (0.0) | 58.8 (4.7) | 55.93 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1
  Male | 2 | 1 | 7 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 8 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 1 | 8 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 8 | 11

OUTCOME MEASURES:

1. Primary Outcome: Response
Description: Overall response is defined as the best response (e.g. complete response...) recorded from the start of treatment until disease progression/recurrence. Complete response is the disappearance of all target lesions. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions. Progressive disease is at least a 20% increase in the sum of LD of target lesions since the treatment started or the appearance of new lesion. Stable disease is neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease.
Time Frame: 3 years and 9 months
Population: Pts in Group C had no evaluable disease,response evaluation was not an appropriate endpoint. The purpose of putting such patients in the trial was they were more likely to survive long enough to complete the full sequence of intended vaccinations and permit an immunological/laboratory endpoint evaluation (not as likely for Groups A and B).
Measure: Count of Participants; unit: Participants
Groups:
- Grp A-measurable Metastatic Disease (no Immediate Aldesleukin): Patients who do not need or are ineligible for treatment with interleukin-2 (IL-2) and patients who have previously had IL-2 therapy.
  A3 FGF-5 (Fibroblast growth factor 5): 172-176/217-220 peptide - two 1 ml injections in the anterior thigh deep subcutaneous tissue within 2c of each other.
  Because patients in Group C had no evaluable disease, response evaluation was not an appropriate endpoint. The purpose of putting such patients in the trial was they were more likely to survive long enough to complete the full sequence of intended vaccinations and permit an immunological/laboratory endpoint evaluation (not as likely for Groups A and B).
Arm/Group | Grp A-measurable Metastatic Disease (no Immediate Aldesleukin) | Grp B - Measurable Metastatic Disease That Require Aldesleukin
Number analyzed (Participants) | 2 | 1
Participants
  Complete response | 0 | 0
  Partial Response | 0 | 0
  Progressive disease | 2 | 1
  Stable disease | 0 | 0
  Not evaluable | 0 | 0

2. Primary Outcome: Count of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events, see the adverse event module.
Time Frame: 47 months
Measure: Count of Participants; unit: Participants
Arm/Group | Grp A-measurable Metastatic Disease (no Immediate Aldesleukin) | Grp B - Measurable Metastatic Disease That Require Aldesleukin | Grp C - High-risk Loco-regional Disease
Number analyzed (Participants) | 2 | 1 | 8
Participants | 2 | 1 | 8

3. Primary Outcome: Immunologic Response to Peptide Vaccination Pre and Post Vaccination
Description: FGF-5 specific CTL (cytotoxic T lymphocytes) may be tested by cytokine release assay or ELISPOT (enzyme linked immunosorbent spot) assay using tumor, FGF-5 transfected or peptide-loaded target cells and compared to pre-treatment peripheral blood mononuclear cells (PBMC) to determine immune response to vaccination. In the assays, differences of 2-3 fold are indicative of true biologic difference.Due to text data entry field limitations, Pre vaccination and post vaccination will be shown in the results as Pre V and Post V, respectively. Patients entered in Group A did not complete sufficient vaccinations to permit immunological evaluation and in Group B, the co-administration of IL-2 is known to corrupt immunological evaluation (so only clinical responses are valid). Expanding information on cancer vaccines in general as wells as preliminary information from this trial on FGF-5 as a vaccine target both served to render the enrollment of additional patients to this trial obsolete.
Time Frame: 24 hours
Population: "1 uM A3 culture vs tranfectant" means "Immune cells cultured with the concentration of 1 uM of the A3 peptide were tested against [with] target cells into which the FGF-5 target gene was inserted [transfected with] and the release of interferon is measured to detect immune recognition".Documentation was only available for the 4 patients.
Measure: Number; unit: pg/ml/24 hrs
Arm/Group | Grp C - High-risk Loco-regional Disease
Number analyzed (Participants) | 4
pg/ml/24 hrs
  Pre V0 A3 pt #1 1µM culture A3/gp100 | 0
  Pre V0 A3 pt #1 1µM culture A3/FGF-5 | 0
  Post V1 A3 pt #1 1µM culture A3/gp100 | 0
  Post V1 A3 pt #1 1µM culture A3/FGF-5 | 1680
  Post V1 A3 pt #1 0.1µM culture A3/FGF-5 | 2620
  Post V1 A3 pt #1 0.01µM culture A3/FGF5 | 4760
  Post V2 A3 pt #1 1µM culture A3/gp100 | 0
  Post V2 A3 pt #1 1µM culture A3/FGF-5 | 826
  Post V2 A3 pt #1 0.1µM culture A3/FGF-5 | 891
  Post V2 A3 pt #1 0.01µM culture A3/FGF5 | 668
  Pre V0 A3 pt #2 1µM culture A3/gp100 | 6
  Pre V0 A3 pt #2 1µM culture A3/FGF-5 | 30
  Pre V0 A3 pt #2FGF-5 culture vs transfectant | 41
  Post V1 A3 pt #2 1µM culture A3/gp100 | 10
  Post V1 A3 pt #2 1µM culture A3/FGF-5 | 258
  Post V1 A3 pt #2FGF-5 culture vs transfectant | 170
  Post V2 A3 pt #2 1µM culture A3/gp100 | 52
  Post V2 A3 pt #2 0.1µM culture A3/FGF-5 | 1424
  Post V2 A3 pt #2FGF-5 culture vs transfectant | 1000
  Pre V0 A3 pt #3 1µM culture A3/gp100 | 2
  Pre V0 A3 pt #3 1µM culture A3/FGF-5 | 1
  Pre V0 A3 pt #3FGF-5 culture vs transfectant | 2
  Post V1 A3 pt #3 1µM culture A3/gp100 | 2
  Post V1 A3 pt #3 1µM culture A3/FGF-5 | 4
  Post V1 A3 pt #3FGF-5 culture vs transfectant | 2
  Post V2 A3 pt #3 1µM culture A3/gp100 | 3
  Post V2 A3 pt #3 0.1µM culture A3/FGF-5 | 9
  Post V2 A3 pt #3FGF-5 culture vs transfectant | 5
  Pre V0 A2 pt #4 1µM culture A2/gp100 | 8
  Pre V0 A2 pt #4 1µM culture A2/FGF-5 | 1
  Pre V0 A2 pt #4FGF-5 culture vs transfectant | 2
  Post V1 A2 pt #4 1µM culture A2/gp100 | 2
  Post V1 A2 pt #4 1µM culture A2/FGF-5 | 68
  Post V1 A2 pt #4FGF-5 culture vs transfectant | 206

ADVERSE EVENTS:
Time Frame: 47 months
Arm/Group | Grp A-measurable Metastatic Disease (no Immediate Aldesleukin) | Grp B - Measurable Metastatic Disease That Require Aldesleukin | Grp C - High-risk Loco-regional Disease
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/1 | 1/8
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Grp A-measurable Metastatic Disease (no Immediate Aldesleukin) (N=2) | Grp B - Measurable Metastatic Disease That Require Aldesleukin (N=1) | Grp C - High-risk Loco-regional Disease (N=8)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Grp A-measurable Metastatic Disease (no Immediate Aldesleukin) (N=2) | Grp B - Measurable Metastatic Disease That Require Aldesleukin (N=1) | Grp C - High-risk Loco-regional Disease (N=8)
Hemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (aPTT) (Investigations) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (2) | 0 (0) | 1 (1)
Injection site reaction (Injury, poisoning and procedural complications) | 2 (5) | 1 (4) | 8 (83)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Metabolism and nutrition disorders) | 1 (2) | 1 (4) | 0 (0)
Serum magnesium increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Metabolism and nutrition disorders) | 2 (3) | 1 (3) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
lymphocyte count decreased (Investigations) | 0 (0) | 1 (4) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis infective (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Bilirubin increased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
serum calcium decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No